CLINICAL TRIAL: NCT05183854
Title: Phase II Study of the Efficacy of the Pneumococcal Pneumonia Vaccine Series in Patients With Chronic Lymphocytic Leukemia Associated Immunodeficiency (PROTECT CLL)
Brief Title: Pneumococcal Pneumonia Vaccine Series (PCV20 and PPSV23) in Patients With Chronic Lymphocytic Leukemia Associated Immunodeficiency, PROTECT CLL Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI145280; NCI-2021-13373 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI145280 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (PCV20, PPSV23) (Experimental): Patients receive pneumococcal 20-valent conjugate vaccine IM on day 1. PnumoVax23 will be given as an intramuscular injection on Visit 2 (approximately Day 75)
  Interventions: Biological: Pneumococcal 20-valent Conjugate Vaccine; Biological: Pneumococcal Polyvalent Vaccine; Other: Questionnaire Administration
- Arm II (PCV20, PPPSV23) (Experimental): Patients who have received or are receiving venetoclax therapy, receive pneumococcal 20-valent conjugate vaccine IM at study visit 1 and pneumococcal polyvalent vaccine IM at study visit 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pneumococcal 20-valent Conjugate Vaccine; Biological: Pneumococcal Polyvalent Vaccine; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Pneumococcal 20-valent Conjugate Vaccine — Given IM
  Other Names: PCV 20; PCV 20 Vaccine; Prevnar 20
Biological: Pneumococcal Polyvalent Vaccine — Given IM
  Other Names: PCV 23; Pneumococcal 23-valent Polysaccharide Vaccine; Pneumococcal Polysaccharide Vaccine; Pneumococcal Vaccine Polyvalent; Pneumovax 23; Pnu-Imune 23; PPSV; PPSV23; PPSV23 Vaccine
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests whether the pneumococcal pneumonia vaccine series (PCV20 and PPSV23) works to mount an effective immune response in patients with chronic lymphocytic leukemia. PCV20 and PPSV23 are both vaccines that protect against bacteria that cause pneumococcal disease. Giving these vaccinations as series may make a stronger immune response and prevent against pneumococcal infections in patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the proportion of chronic lymphocytic leukemia (CLL) patients who mount an effective immune response to streptococcus pneumonia after receiving both pneumococcal 20-valent conjugate vaccine (PCV20) and pneumococcal polyvalent vaccine (PPSV23) vaccinations. (Primary Analysis)

SECONDARY OBJECTIVES:

I. To improve the immunoglobulin levels and decrease the incidence of pneumonia in patients with CLL-associated immunodeficiency. (Primary Analysis) II. To evaluate the rate of decreased pneumonia as assessed by an immune response to streptococcus (S.) pneumoniae after PCV20 and PPSV23 series versus PCV20 alone. (Primary Analysis) III. To investigate the immune response to individual S. pneumoniae serotypes included in both the PCV20 and PPSV23 vaccinations. (Primary Analysis) IV. Evaluate the length of time an effective immune response is maintained, and if the recommendation of 5 years is adequate for CLL patients. (Primary Analysis)

EXPLORATORY OBJECTIVES:

I. Assess rate of pneumonia in CLL patients based on therapeutic strategy (i.e., BTKi, venetoclax, chemo-immunotherapy).

II. To evaluate the number of venetoclax treated CLL patients who mount an effective immune response to S. pneumoniae 30 days following both PCV20 and PPSV23 vaccinations. (Pilot Arm)

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (PRIMARY ARM): Patients receive pneumococcal 20-valent conjugate vaccine intramuscularly (IM) on day 1 and pneumococcal polyvalent vaccine IM on day 60 in the absence of disease progression or unacceptable toxicity.

ARM II (PILOT ARM): Patients who have received or are receiving venetoclax therapy, receive pneumococcal 20-valent conjugate vaccine IM on day 1 and pneumococcal polyvalent vaccine IM on day 60 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 90 days and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* NAIVE COHORT: Subjects must have a confirmed diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) (collectively referred to as CLL throughout) according to the 2018 International Workshop on CLL.
* NAIVE COHORT: Male or female subject aged >= 18 years.
* NAIVE COHORT: Subjects must not have received prior therapy for CLL.
* VENETOCLAX-TREATMENT COHORT: Subjects must have a confirmed diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) (collectively referred to as CLL throughout) according to the 2018 International Workshop on CLL.
* VENETOCLAX-TREATMENT COHORT: Subjects must have received venetoclax (any dose) for at least 12 months with the last dose =< 12 months prior to registration.

Exclusion Criteria:

* Subjects who have experienced a severe allergic reaction to prior pneumococcal vaccination.
* Subjects who have received a PCV13 or PCV20 pneumococcal vaccination in the last five years.
* If they have received PPSV23 in ≥ 1 year and no other pneumococcal vaccine they may be included.
* Active infection requiring systemic antibiotic therapy.
* Current or prior use of immunosuppressive medication within 14 days of cycle one day one, EXCEPT for the following permitted steroids:

  * Intranasal, inhaled, topical steroids, eye drops or local steroid injection (e.g., intra-articular injection);
  * Systemic corticosteroids at physiologic doses =< 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).
* Concurrent illness or condition, which, in the opinion of the treating investigator, would negatively impact the subject's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2028-01-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve the protocol defined change in antibody titers | At 30 and 90 days post-PCV20 vaccination
  Will examine the proportion of patients who achieve the protocol defined change in antibody titers from baseline in at least 10 of 19 S.pneumoniae serotypes shared between pneumococcal 20-valent conjugate vaccine (PCV20) and pneumococcal polyvalent vaccine (PPSV23) at Study Visit 2 and 3. The observed proportion and an exact 95% binomial confidence interval will be reported. A one sample exact binomial test will be performed at one-sided alpha = 0.05. The null hypothesis is that the proportion is 50% or lower.

SECONDARY OUTCOMES:
Proportion of patients who have a two-fold increase of immunoglobulin levels | Up to 5 years post- PPSV23 vaccination
  Will examine the proportion of patients who have a two-fold increase of immunoglobulin levels from baseline at Study Visit 2 and 3 and do not develop pneumonia within five years post-PPSV23 vaccination. The observed proportion and an exact 95% binomial confidence interval will be reported.
Proportion of vaccinated patients who have a two-fold increase in at least 10 of 19 S. pneumonia serotypes shared between PCV20 and PPSV23 vaccines | Up to 5 years post PPSV23 vaccination
  Will examine the proportion of vaccinated patients who have a two-fold increase in at least 10 of 19 S. pneumonia serotypes shared between PCV20 and PPSV23 vaccines and do not develop pneumonia within five years post PPSV23 vaccination. The observed proportion and an exact 95% binomial confidence interval will be reported.
Proportion of patients who have a two-fold increase in antibody titers to an individual serotype vaccination | At 30 and 90 days post-PCV20 vaccination
  Will examine the proportion of patients who have a two-fold increase in antibody titers to an individual serotype at Study Visit 2 and 3 post PPCV20 vaccination. The observed proportion and 95% exact binomial confidence intervals will be reported for each serotype.
Proportion of patients who maintain adequate immune response | Up to 5 years post PPSV23 vaccination
  Will examine the proportion of patients who maintain adequate immune response, defined as two-fold increase in antibody titers from baseline in 10/19 of S. pneumoniae serotypes, from PPSV23 vaccination to time of last follow-up at 5 years. Kaplan-Meier methods will be used to analyze time-to-pneumonia from baseline until five years after PPSV23 vaccination.

OTHER OUTCOMES:
Number of patients that contract pneumonia | Up to 5 years post PPSV23 vaccination
  Kaplan-Meier methods will be used to analyze time-to-pneumonia from baseline until five years after study entry, stratified by therapeutic strategy.
Proportion of venetoclax treated chronic lymphocytic leukemia (CLL) patients who achieve a two-fold increase in antibody titers | At 30 and 90 days post PCV20 vaccination
  Will examine the proportion of Venetoclax treated CLL patients who achieve a two-fold increase in antibody titers from baseline in at least 10 of 19 S. pneumonia serotypes shared between PCV20 and PPSV23 vaccines at Study Visit 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ermann, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No